CLINICAL TRIAL: NCT03266068
Title: Epidemiology and Pathophysiology of Post-Infectious Functional GI Disorders
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Madhusudan (Madhu) Grover, MBBS, Assistant Professor of Medicine, Mayo Clinic
Other Study IDs: 12-006529; K23DK103911 (NIH); P30DK084567 (NIH); UL1TR000135 (NIH)
Record Dates: First submitted 2017-07-05; First posted 2017-08-29 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Campylobacter Infections; Irritable Bowel Syndrome
MeSH Terms: conditions — Campylobacter Infections; Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, stool, and tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Post Infectious IBS Case: Subjects who have suffered from acute bacterial gastroenteritis within last two years and have developed some symptoms that might be suggestive of post-infectious irritable bowel syndrome (IBS). Subjects will receive a DNA analysis of blood sample, flexible sigmoidoscopy with colonic biopsies, small bowel and colonic gastrointestinal permeability, and stool sample analysis.
  Interventions: Genetic: DNA Analysis of Blood Sample; Procedure: Flexible sigmoidoscopy with colonic biopsies; Procedure: Small bowel and colonic gastrointestinal permeability; Diagnostic Test: Stool sample analysis
- Post Infectious with no IBS Control: Subjects who have suffered from acute bacterial gastroenteritis within last two years and have not developed symptoms suggestive of post-infectious irritable bowel syndrome (IBS). Subjects will receive a DNA analysis of blood sample, flexible sigmoidoscopy with colonic biopsies, small bowel and colonic gastrointestinal permeability, and stool sample analysis.
  Interventions: Genetic: DNA Analysis of Blood Sample; Procedure: Flexible sigmoidoscopy with colonic biopsies; Procedure: Small bowel and colonic gastrointestinal permeability; Diagnostic Test: Stool sample analysis
- Healthy Control: Healthy volunteers; subjects will receive a DNA analysis of blood sample, flexible sigmoidoscopy with colonic biopsies, small bowel and colonic gastrointestinal permeability, and stool sample analysis.
  Interventions: Genetic: DNA Analysis of Blood Sample; Procedure: Flexible sigmoidoscopy with colonic biopsies; Procedure: Small bowel and colonic gastrointestinal permeability; Diagnostic Test: Stool sample analysis

INTERVENTIONS:
Genetic: DNA Analysis of Blood Sample — DNA analysis of the genes possibly involved in IBS.
Procedure: Flexible sigmoidoscopy with colonic biopsies — Endoscopy of the subject's lower colon in which biopsies of the lining of the colon will be taken.
Procedure: Small bowel and colonic gastrointestinal permeability — A validated scintigraphic method to measure gastric, small bowel and colonic transit will be used.
Diagnostic Test: Stool sample analysis — Stool samples will be used to extract supernatants. These supernatants will be studied in using chamber set-up to determine barrier effects on T84 monolayers.

SUMMARY:
Some people develop chronic abdominal pain with diarrhea or constipation after an episode of acute bacterial gastroenteritis. These symptoms can be consistent with post-infectious irritable bowel syndrome (IBS) and can last long after the acute infection is over. The exact reason why certain individuals develop these symptoms whereas others don't is not exactly clear.

The researchers are studying changes in gastrointestinal permeability (movement of contents across the lining of the intestine) and transit (movement of food through the gastrointestinal tract). The researchers are also studying if there are any genetic risk factors that are associated with development of this disorder.

DETAILED DESCRIPTION:
The Centers for Disease Control and prevention (CDC) estimates that each year roughly 1 in 6 Americans (or 48 million people) contact food-borne illnesses. The CDC also estimates that between 20 and 40% of individuals traveling to a developing country get traveler's diarrhea. There is morbidity from these illnesses, even after the acute episode is over. Thus, up to a third of patients suffering from acute infectious gastroenteritis (IGE), most often resulting from a food-borne outbreak or travel develop chronic gastrointestinal (GI) illnesses such as irritable bowel syndrome (IBS). In addition, recent studies are suggesting that military personnel who suffered from IGE during deployment are more likely to suffer from IBS post-deployment. This disorder has been described as post-infectious IBS (PI-IBS).

Individuals with PI-IBS suffer from recurrent, debilitating abdominal pain and altered bowel function (diarrhea and/or constipation) and symptoms can be present for over 8 years after the acute IGE episode is over. It is estimated that up to 15% of the United States population suffers from IBS. This disorder creates significant impact on patient's daily functioning, overall quality of life and causes loss of work productivity. Despite the impact of this illness, treatment options for IBS have limited success, with a significant unmet need. Lack of understanding of underlying pathophysiological mechanisms has hampered development of effective treatment. More studies are required to enhance understanding of this disorder. Development of PI-IBS after an episode of acute IGE serves as a unique model to study risk-factors and mechanisms underlying PI-IBS and IBS in general. The researchers propose to study the epidemiological risk factors and pathophysiological mechanisms involved in the development of IBS among individuals suffering from episodes of acute IGE in the community.

Pathophysiology of IBS includes abnormalities of GI motility, sensation, mucosal defense, immune function and psychosocial factors. The researchers propose to investigate overall risk and patient demographic, pathogen and illness related characteristics as predictors for development of PI-IBS among patients who had suffered from acute IGE. In addition, the researchers want to determine pathophysiological mechanisms leading to the development of this disorder.

In order to achieve these goals, the researchers propose to establish collaboration with the Minnesota Department of Health (MDH) which conducts active surveillance for bacterial and parasitic cases of acute IGE and other reportable illnesses in Minnesota, as part of the mandate to detecting outbreaks and prioritize control efforts. We plan to establish retrospective and prospective cohorts in this proposal. A randomly selected sub-set of these patients will be invited to Mayo Clinic for detailed investigations including assessment of GI motility, permeability, endoscopic examination for colon biopsies, and diverse blood and stool assays using techniques that are all validated to provide information about the mechanism of PI-IBS. The researchers will also investigate variations in the barrier function pathway genes in tissues of PI-IBS patients and to understand the contribution of these genetic variations in immune activation and control of barrier function to increased susceptibility to PI-IBS.

ELIGIBILITY:
Post Infectious IBS Cases Inclusion Criteria:

1. IBS by Rome III criteria
2. No abdominal surgery (except hernia, C-section, hysterectomy, appendectomy and cholecystectomy)

Post Infectious with no IBS Controls Inclusion Criteria:

1. No IBS by Rome III criteria
2. No abdominal surgery (except hernia, C-section, hysterectomy, appendectomy and cholecystectomy)

Post Infectious IBS Cases and Post Infectious with no IBS Controls Exclusion Criteria:

1. Prior history of IBS or inflammatory bowel disease (IBD) (Crohn's disease or ulcerative colitis), microscopic colitis or celiac disease
2. Ingestion of artificial sweeteners such as sucralose, aspartame, lactulose or mannitol 2 days before the study begins, e.g., foods to be avoided are sugarless gums or mints and diet soda
3. Ingestion of any prescription, over the counter, or herbal medications which can affect gastrointestinal transit 7 days before study begins

   1. Any treatment specifically taken for IBS, including loperamide, cholestyramine, alosetron
   2. Drugs with a known pharmacological activity at serotonin type 4 (5-HT4), serotonin receptor 2B (5-HT2b) or 5-HT3 receptors (e.g, tegaserod, ondansetron, tropisetron, granisetron, dolasetron, mirtazapine)
   3. All narcotics (e.g, codeine, morphine, and propoxyphene, either alone or in combination)
   4. Anti-cholinergic agents (e.g, dicyclomine, hyoscyamine, propantheline)
   5. Ultram
   6. GI preparations

      * Anti-nausea agents (e.g, trimethobenzamide, promethazine, prochlorperazine, dimenhydrinate, hydroxyzine)
      * Osmotic laxative agents (e.g, lactulose, sorbitol or polyethylene glycol (PEG) solutions as Miralax and Glycolax)
      * Prokinetic agents (e.g, cisapride, metoclopramide, itopride, domperidone)
   7. Antimuscarinics
   8. Peppermint oil
   9. Systemic antibiotics, rifaximin, metronidazole
4. Any females who are pregnant or trying to become pregnant (due to radiation exposure)
5. Bleeding disorders or medications that increase risk of bleeding from mucosal biopsies

Healthy Control Inclusion Criteria:

1. No abdominal surgery (except hernia, C-section, hysterectomy, appendectomy and cholecystectomy)
2. No history of acute gastroenteritis, food-poisoning or travel related diarrhea within last 2 years.

Healthy Control Exclusion Criteria:

1. Prior history of IBS or IBD (Crohn's disease or ulcerative colitis), microscopic colitis or celiac disease
2. Ingestion of artificial sweeteners such as sucralose, aspartame, lactulose or mannitol 2 days before the study begins, e.g., foods to be avoided are sugarless gums or mints and diet soda
3. Ingestion of any prescription, over the counter, or herbal medications which can affect gastrointestinal transit 7 days before study begins

   1. Any treatment specifically taken for IBS, including loperamide, cholestyramine, alosetron
   2. Drugs with a known pharmacological activity at 5-HT4, 5-HT2b or 5-HT3 receptors (e.g, tegaserod, ondansetron, tropisetron, granisetron, dolasetron, mirtazapine)
   3. All narcotics (e.g, codeine, morphine, and propoxyphene, either alone or in combination)
   4. Anti-cholinergic agents (e.g, dicyclomine, hyoscyamine, propantheline)
   5. Ultram
   6. GI preparations

      * Anti-nausea agents (e.g, trimethobenzamide, promethazine, prochlorperazine, dimenhydrinate, hydroxyzine)
      * Osmotic laxative agents (e.g, lactulose, sorbitol or PEG solutions as Miralax and Glycolax)
      * Prokinetic agents (e.g, cisapride, metoclopramide, itopride, domperidone)
   7. Antimuscarinics
   8. Peppermint oil
   9. Systemic antibiotics, rifaximin, metronidazole
4. Any females who are pregnant or trying to become pregnant (due to radiation exposure)
5. Bleeding disorders or medications that increase risk of bleeding from mucosal biopsies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Post Infectious IBS Cases Post Infectious with no IBS Controls Healthy Volunteer Controls
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Colonic geometric center at 24 hours | 24 hours
  The scintigraphic method is used to measure colonic transit. An isotope is adsorbed on activated charcoal particles and delivered to the colon in a delayed release capsule. Anterior and posterior gamma images are taken hourly. The geometric center (GC) is the weighted average of counts in the different colonic regions. The scale ranges from 1 to 5; a high GC implies faster colonic transit, a GC of 1 implies all isotope is in the ascending colon, and a GC of 5 implies all isotope is in the stool.

CONTACTS AND LOCATIONS:
Overall Officials: Madhusudan Grover, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials